CLINICAL TRIAL: NCT04232033
Title: The Physiological Effects of FGF21 on Alcohol Preference and Glucose Metabolism in Healthy Men
Brief Title: The Physiological Effects of FGF21 on Alcohol Preference and Glucose Metabolism
Acronym: AlcoPref
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: H-19068397
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Fibroblast Growth Factor 21; Tast Perference
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibroblast growth factor 21 infusion (Active Comparator): Fibroblast growth factor 21 infusion
  Interventions: Other: Fibroblast growth factor 21 infusion
- Placebo infusion (saline) (Placebo Comparator): Saline infusion
  Interventions: Other: Placebo infusion (saline)

INTERVENTIONS:
Other: Fibroblast growth factor 21 infusion — Infusion of Fibroblast growth factor 21
  Arms: Fibroblast growth factor 21 infusion
Other: Placebo infusion (saline) — Infusion of Saline
  Arms: Placebo infusion (saline)

SUMMARY:
The primary objective is to evaluate taste preferences for alcohol during an intravenous infusion of the naturally occurring hormone fibroblast growth factor-21 (FGF21) and placebo (i.e. saline), respectively, in 20 healthy subjects. Secondary endpoints are to evaluate the effects of exogenous FGF21 (compared to placebo) on resting energy expenditure, preference for salt, sour and bitter taste qualities, sensations of hunger, thirst, appetite, satiety, headache and nausea, and makers of glucose metabolism (e.g. plasma/serum concentrations of glucose, C-peptide, insulin and glucagon).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Caucasian male
* Body mass index between 19 and 27 kg/m2
* Normal haemoglobin and normal glycated haemoglobin A1c (HbA1c) (< 42 mmol/mol)
* Weekly alcohol intake of less than 14 units of alcohol (1 unit = 12 g ethanol)

Exclusion Criteria:

* Liver diseases evaluated by plasma alanine aminotransferase (ALAT) > 3 × normal level or an International Normalized Ratio (INR) below normal values
* Diabetes mellitus
* Nephropathy
* First-degree relatives with diabetes and/or liver diseases and/or alcohol use disorder
* Other diseases the investigator finds disruptive for participation in the study

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Alcohol preference (How much do you want to drink alcohol?) | 1 year
  Evaluated by Visual analogue scale from "not at all" to "more than ever"

SECONDARY OUTCOMES:
Plasma glucose concentration | 1 year
  Plasma glucose concentration
Serum insulin concentration | 1 year
  Serum insulin concentration
Plasma fibroblast growth factor-21 concentration | 1 year
  Plasma fibroblast growth factor-21 concentration
Serum C-peptide concentration | 1 year
  Serum C-peptide concentration
Plasma glucagon concentration | 1 year
  Serum C-peptide concentration
Plasma lipid profile | 1 year
  Plasma concentrations of triglycerides, total cholesterol, free fatty acids
Plasma insulin-like growth factor 1 concentration | 1 year
  Plasma insulin-like growth factor 1 concentration
Plasma bone marker concentration | 1 year
  Plasma concentrations of the bone markers carboxy-terminal collagen crosslink and procollagen type 1 N-terminal propeptide
Resting energy expenditure | 1 year
  Evaluated by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Amalie R Lanng, Dr., Principal Investigator — Center for Clinical Metabolic Research, Gentofte Hospital
Locations (1):
- Amalie R Lanng, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.